CLINICAL TRIAL: NCT00893373
Title: A Double-blind, Placebo-controlled, Randomized, Multicenter Phase-II Trial to Assess the Efficacy of Sorafenib Added to Standard Primary Therapy in Patients With Newly Diagnosed AML ≤60 Years of Age
Brief Title: Study Evaluating Sorafenib Added to Standard Primary Therapy in Patients With Newly Diagnosed Acute Myeloid Leukemia Less Than 60 Years of Age
Acronym: SORAML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUD-SORAML-034
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: AML; sorafenib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Experimental): Induction, Consolidation and Maintenance plus Sorafenib 2x 400 mg/d
  Interventions: Drug: sorafenib
- Placebo (Placebo Comparator): Induction, Consolidation and Maintenance plus Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sorafenib — Standard AML chemotherapy plus sorafenib 400 mg BID
  Other Names: nexavar
  Arms: Sorafenib
Drug: placebo — Standard AML chemotherapy plus placebo
  Arms: Placebo

SUMMARY:
Sorafenib is a multikinase inhibitor which is acting on various cellular pathways involved in the genesis of acute myeloid leukemia (AML). Sorafenib is therefore a promising candidate for improvement of chemotherapy results in AML. This clinical trial evaluates the efficacy of sorafenib added to standard chemotherapy for AML in patients between 18 and 60 years of age. Patients are randomised to receive either sorafenib capsules or placebo in addition to their chemotherapy. The placebo and the sorafenib group will be compared regarding event-free survival and other clinical outcomes. An event is either treatment failure or relapse or death. According to the study hypothesis, the sorafenib group will have less events than the placebo group.

ELIGIBILITY:
Inclusion criteria:

* Patients with newly diagnosed AML (except APL) according to the FAB and WHO classification, including AML evolving from MDS or other hematologic diseases and AML after previous cytotoxic therapy or radiation (secondary AML)
* Bone marrow aspirate or biopsy must contain ≥ 20% blasts of all nucleated cells or differential blood count must contain ≥ 20% blasts. In AML FAB M6 ≥ 30% of nonerythroid cells in the bone marrow must be leukemic blasts. In AML defined by cytogenetic aberrations, the proportion of blasts may be < 20%.
* Age ≥ 18 and ≤ 60 years
* Informed consent, personally signed and dated to participate in the study
* ECOG performance status of 0-1
* Life expectancy of at least 12 weeks
* Adequate liver and renal function as assessed by laboratory requirements to be conducted within 7 days prior to Screening

Exclusion criteria:

* Patients who are not eligible for standard chemotherapy as per discretion of the treating physician
* Central nervous system manifestation of AML
* Cardiac disease: heart failure NYHA III or IV; unstable coronary artery disease (MI more than 6 months prior to study entry is permitted); serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Chronically impaired renal function (creatinine clearance < 30 ml/min) (Cockcroft-Gault formula)
* Patients undergoing renal dialysis
* Chronic pulmonary disease with relevant hypoxia
* Known HIV and/or hepatitis C infection
* Evidence or history of severe non-leukemia associated bleeding diathesis or coagulopathy
* Evidence or recent history of CNS disease, including primary or metastatic brain tumors, seizure disorders
* Resting blood pressure (BP) consistently higher than systolic 160 mmHg and/or diastolic 95 mmHg
* Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance of the protocol
* Patients with major surgery, open biopsy or significant traumatic injury within 4 weeks of start of first dose
* Serious, non-healing wound, ulcer or bone fracture
* Uncontrolled active infection > Grade 2 NCI-CTC version 3.0
* Concurrent malignancies other than AML
* History of organ allograft
* Allergy to study medication or excipients in study medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 36 months

SECONDARY OUTCOMES:
Overall survival | 36 months
Rate of complete remissions | 12 weeks
Toxicity | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Ehninger, Prof, MD, Principal Investigator — University Hospital Dresden
Locations (9):
- Germany (9):
  - Sozialstiftung Bamberg Klinikum am Bruderwald, Bamberg
  - Klinikum Bayreuth, Bayreuth
  - Charite Campus Benjamin Franklin, Berlin
  - Ev. Diakonie-Krankenhaus gGmbH Bremen, Bremen
  - University Hospital Dresden, Dresden
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Agaplesion Diakoniekrankenhaus Rotenburg, Rotenburg (Wümme)
  - Robert-Bosch-Krankenhaus, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kunadt D, Stasik S, Metzeler KH, Rollig C, Schliemann C, Greif PA, Spiekermann K, Rothenberg-Thurley M, Krug U, Braess J, Kramer A, Hochhaus A, Scholl S, Hilgendorf I, Brummendorf TH, Jost E, Steffen B, Bug G, Einsele H, Gorlich D, Sauerland C, Schafer-Eckart K, Krause SW, Hanel M, Hanoun M, Kaufmann M, Wormann B, Kramer M, Sockel K, Egger-Heidrich K, Herold T, Ehninger G, Burchert A, Platzbecker U, Berdel WE, Muller-Tidow C, Hiddemann W, Serve H, Stelljes M, Baldus CD, Neubauer A, Schetelig J, Thiede C, Bornhauser M, Middeke JM, Stolzel F; A. M. L. Cooperative Group (AMLCG), Study Alliance Leukemia (SAL). Impact of IDH1 and IDH2 mutational subgroups in AML patients after allogeneic stem cell transplantation. J Hematol Oncol. 2022 Sep 5;15(1):126. doi: 10.1186/s13045-022-01339-8. PMID 36064577
- [Derived] Rollig C, Serve H, Huttmann A, Noppeney R, Muller-Tidow C, Krug U, Baldus CD, Brandts CH, Kunzmann V, Einsele H, Kramer A, Schafer-Eckart K, Neubauer A, Burchert A, Giagounidis A, Krause SW, Mackensen A, Aulitzky W, Herbst R, Hanel M, Kiani A, Frickhofen N, Kullmer J, Kaiser U, Link H, Geer T, Reichle A, Junghanss C, Repp R, Heits F, Durk H, Hase J, Klut IM, Illmer T, Bornhauser M, Schaich M, Parmentier S, Gorner M, Thiede C, von Bonin M, Schetelig J, Kramer M, Berdel WE, Ehninger G; Study Alliance Leukaemia. Addition of sorafenib versus placebo to standard therapy in patients aged 60 years or younger with newly diagnosed acute myeloid leukaemia (SORAML): a multicentre, phase 2, randomised controlled trial. Lancet Oncol. 2015 Dec;16(16):1691-9. doi: 10.1016/S1470-2045(15)00362-9. Epub 2015 Nov 6. PMID 26549589
- [Derived] Herold T, Metzeler KH, Vosberg S, Hartmann L, Rollig C, Stolzel F, Schneider S, Hubmann M, Zellmeier E, Ksienzyk B, Jurinovic V, Pasalic Z, Kakadia PM, Dufour A, Graf A, Krebs S, Blum H, Sauerland MC, Buchner T, Berdel WE, Woermann BJ, Bornhauser M, Ehninger G, Mansmann U, Hiddemann W, Bohlander SK, Spiekermann K, Greif PA. Isolated trisomy 13 defines a homogeneous AML subgroup with high frequency of mutations in spliceosome genes and poor prognosis. Blood. 2014 Aug 21;124(8):1304-11. doi: 10.1182/blood-2013-12-540716. Epub 2014 Jun 12. PMID 24923295
- See also: SAL - Study Alliance Leukemia — http://www.sal-aml.org